CLINICAL TRIAL: NCT01993862
Title: Safety and Cost Effectiveness of Same Day Discharge After Implantable Cardioverter-Defibrillator Implant Versus Next Day Discharge
Brief Title: Same Day Discharge (SDD) After Implantable Cardioverter Defibrillator (ICD) Implant
Acronym: SDD for ICD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 40009529/B
Record Dates: First submitted 2013-11-19; First posted 2013-11-25 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Heart Failure; Coronary Artery Disease
MeSH Terms: conditions — Heart Failure; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Next Day Discharge (No Intervention): The patient will have a 23 hour standard of care observational stay in the hospital after an implantable cardioverter defibrillator implant procedure.
- Same Day Discharge (Active Comparator): The patient will be discharged from the hospital the same evening after an implantable cardioverter defibrillator implant procedure. Follow up after surgery will be done via remote device follow up (1) on the day of discharge and (2) 24 hours after surgery.
  Interventions: Other: Same Day Discharge

INTERVENTIONS:
Other: Same Day Discharge — Patients will send device data remotely to their physician on the day of discharge from the hospital and again 24 hours after discharge from the hospital.
  Arms: Same Day Discharge

SUMMARY:
The purpose of this study is to determine whether it is safe to send patients home from the hospital on the same day following an implantable cardioverter defibrillator (ICD) implant.

DETAILED DESCRIPTION:
SDD for ICD is a prospective, randomized, multi-center study designed to show that SDD is safe in a defined patient population receiving an ICD implant and that this approach can be more cost effective for the hospital than the current NDD approach. Safety is to be demonstrated by showing that postoperative complications do not occur at a higher rate in the SDD group of patients when compared to the NDD group. Cost effectiveness is to be demonstrated by comparing health care utilization between the SDD and NDD groups for the first week post implantation. Patients who were implanted with a St. Jude Medical single or dual chamber ICD for primary prevention and who met all inclusion and exclusion criteria may be enrolled in the study. Patients areconsidered enrolled at the point of randomization.

Randomization is assigned in a 1:1 ratio between the NDD group and the SDD group. Patients will undergo study evaluations after implant, pre-discharge, 1-week and 6 months post implant.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a St Jude Medical device that is compatible with Merlin.net (remote monitoring)
* Patient is receiving an implantable cardioverter defibrillator for primary prevention
* Patient lives within 50 miles of an emergency room or 24 hour urgent care
* Patient is able to sign informed consent

Exclusion Criteria:

* Patient experiences a complication during or 4 hours after implantable cardioverter defibrillator procedure
* Physician elects to keep the patient in over night due to a change in medical condition or a pre-existing condition that requires administration of continuous blood thinners
* Physician is unable to program the implantable cardioverter defibrillator to collect all required information remotely from device
* Patient is pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2014-03-17 (Actual); Primary Completion 2016-08-05 (Actual); Study Completion 2016-08-12 (Actual)

PRIMARY OUTCOMES:
Complication rate at 1 week after an implantable cardioverter defibrillator implant | 1 week

SECONDARY OUTCOMES:
Cost savings per patient | 1 week
Complication rate at 6 months after an implantable cardioverter defibrillator implant | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Indrajit Choudhuri, MD, Principal Investigator — University of Wisconsin, Madison; Ranjit Suri, MD, Principal Investigator — Heart Rhythm Associates of New York, NY
Locations (28):
- United States (28):
  - Heart Center Research, Huntsville, Alabama
  - Cardiology Associates of Mobile, Mobile, Alabama
  - John C Lincoln North Mountain Hospital, Phoenix, Arizona
  - Chula Vista Cardiac Center, Chula Vista, California
  - Cardiovascular Consultants Heart Center, Fresno, California
  - Stanislaus Cardiology Group, Modesto, California
  - Sutter Medical Center of Santa Rosa, Santa Rosa, California
  - Exempla Rocky Mountain Cardiovascular Associates, Broomfield, Colorado
  - South Denver Cardiology Associates PC, Littleton, Colorado
  - Lakeland Regional Medical Center, Lakeland, Florida
  - Watson Clinic Center, Lakeland, Florida
  - Florida Cardiovascular Specialists, Leesburg, Florida
  - Naples Heart Rhythm Specialists, PA, Naples, Florida
  - Loyola University Medical Center, Maywood, Illinois
  - Chicago Cardiology Institute, Schaumburg, Illinois
  - Ochsner Medical Center, New Orleans, Louisiana
  - Delmarva Heart, Salisbury, Maryland
  - Thoracic Cardiovascular Healthcare Foundation, Lansing, Michigan
  - Great Lakes Heart and Cascular Institute PC, Saint Joseph, Michigan
  - Jackson Heart Clinic, Jackson, Mississippi
  - Missouri Baptist Medical Center, St Louis, Missouri
  - St. Louis Heart and Vascular PC, St Louis, Missouri
  - The New York Hospital Queens, Flushing, New York
  - St. Luke's Hospital - Roosevelt, New York, New York
  - Cary Cardiology, PA, Cary, North Carolina
  - Cardiology Consultants, Johnson City, Tennessee
  - Arrhythmia Associates of South Texas, San Antonio, Texas
  - Aurora Medical Group, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided